CLINICAL TRIAL: NCT06467981
Title: Study of the Indications for Amyloid PET Scans and Their Usefulness in the Management of Patients With Suspected Alzheimer's Disease (AD)
Brief Title: Study of the Indications for Amyloid Positon Emission Tomography (PET) Scans and Their Usefulness for Patients With Suspected Alzheimer's Disease (AD)
Acronym: TEPAmy
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, Investigator coordinator, Central Hospital, Nancy, France
Other Study IDs: 2024PI105
Record Dates: First submitted 2024-06-11; First posted 2024-06-21 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2024-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Retrospective study — The data from the PET request form will be collected in each center for this population of patients who have had an amyloid PET scan with flutemetamol and the results of the PET examination reports will also be provided, all data will be made anonymous.
  Other Names: Filled request form of PET for each patient

SUMMARY:
The recent clinical authorization of amyloid Positon Emission Tomography (PET) in France represents a crucial step for the nuclear medicine community involved in the diagnosis of Alzheimer's disease (AD).

DETAILED DESCRIPTION:
The recent clinical authorization of amyloid Positon Emission Tomography (PET) in France represents a crucial step for the nuclear medicine community involved in the diagnosis of Alzheimer's disease (AD). At the era of Amyloid, Tau, Neurodegeneration (ATN) biomarkers, amyloid PET fills a need in patients with an atypical or mixed clinical presentation, in particular young patients (< 65 years old), when the lumbar puncture is contraindicated or not feasible for technical reasons. Importantly, a negative amyloid PET scan discards the diagnosis of AD. Furthermore, early phase imaging of amyloid PET allows to estimate the perfusion neuronal state, increasing the diagnostic value of such PET radiotracer. Its role could be further developed in routine care for the selection and monitoring of promising disease modifiers therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged = or > 18 years
* Patients who have had an amyloid PET scan with a PET request form including the indications for the examination
* Patient informed via a newsletter and non-opposition to the use of their data for research purposes (research objectives clearly explained in the letters)

Exclusion Criteria:

* Patient opposition to the use of their data for this research

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had a flutemetamol amyloid PET scan with a PET request form including the indications for the examination and who received the information letter on the objectives of the research and who did not object to the use of their data.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Evaluate the indications for Amyloid PET in 7 centers in France to assess the relevance of the examination | 1 day
  Correlation between the request and the recommendations

SECONDARY OUTCOMES:
Evaluate the frequency of positive examinations for the diagnosis of AD | 1 day
  Number of positive PET exam

CONTACTS AND LOCATIONS:
Locations (1):
- Nuclear medicine department, Vandœuvre-lès-Nancy, France